CLINICAL TRIAL: NCT06433388
Title: Perirenal Fats of Chronic Kidney Disease in Patients With Fatty Liver Disease.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Ahmed Ramadan Mohamed, Doctor, Assiut University
Other Study IDs: perirenal fats of ckd
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Diseases; Fatty Liver
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Magnetic Resonance Imaging (MRI) is a non-invasive imaging technology that produces three dimensional detailed anatomical images. Patients will be subjected to MRI scans and imaging of the kidneys and liver

SUMMARY:
Exploring the association of perirenal fat thickness assessed by MRI in CKD patients with FLD.

DETAILED DESCRIPTION:
Fatty liver disease (FLD) is caused by an accumulation of excessive fat in the liver that leads to liver damage. It has been noticed that fatty liver disease affects not only liver diseases but also extra-hepatic organ systems such as the cardiovascular and renal systems. Increasing the prevalence of FLD has a great association with increasing the risk of cardiovascular diseases, chronic kidney diseases, and Type 2 diabetes mellitus. Hypertension, insulin resistance, and abdominal obesity are risk factors that are shared by FLD and CKD. Moreover, patients with CKD have a great prevalence of developing FLD, and CKD incidence is increased by the presence of FLD.

Obesity is one of the most comorbidities over the world, it is related and increase the risk of cardio metabolic disease, as well as it is a strong risk factor for chronic kidney disease (CKD), and the prevalence of both conditions is rising worldwide, Several recent epidemiologic studies have shown that obesity and the metabolic syndrome are independent predictors of CKD. The most common method for defining obesity is based on BMI(weight [kilograms] divided by the square of height [meters]).

previously abdominal fat distribution have been measured by BMI, waist to hip ratio (WHR), OR Waist circumference. Although waist circumference was noted to be a reliable predictor of visceral fat, many interfering factors may also reduce the reliability of WC in estimating abdominal fat deposition, as well as the associated risk for CKD like ageing and normal difference in fat distribution between the two genders. Based on these considerations, we presume that per renal fat thickness measurement by MRI may better reflect the risks commonly associated with increased visceral fat accumulation and particularly those related to renal function impairment.

Chronic kidney disease is defined as impairment or structural damage to kidney or kidney function. It manifested by reduction in estimated glomerular rate (eGFR) for at least 3 months. It presented with proteinuria or albuminuria, hematuria. The best diagnosis by biopsy showing renal impairment, or by imaging ultrasound. CKD associated with morbidity and mortality condition especially in developing countries, so it has been necessary to early detection to prevent CKD progression and associated complications, thus improving patient outcomes and reducing the impact of CKD on health-care resources.

FLD begins with liver lipid accumulation, and marked hepatic fat accumulation is a risk factor for disease progression. Liver biopsy is the golden for diagnosis and assessment of the severity of steatosis and grading of fibrosis, although being invasive and difficult method. Ultrasound and magnetic resonance imaging (MRI) biomarkers of liver fat Gives the advantage diagnose FLD as it is non-invasive imaging biomarkers to diagnose FLD, steatosis , and fibrosis.

Therefore the aim of this study is to determine the independent association of Perirenal fat assessment by MRI with the main markers of kidney function, such as estimated glomerular filtration rate (eGFR), albuminuria as well as with serum urate values on one side, and grading of fibrosis and steatosis in FLD patients on the other side.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old regardless of gender

Exclusion Criteria:

* Other causes of chronic liver diseases (HCV, HBV...).
* End stage renal diseases (GFR<15 ml/min).
* A history of significant alcohol intake (>20 g/day in females and 30 g/day in males).
* Those using medications that can cause fatty liver.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the out-patient clinics of the Internal Medicine Department, Assiut university
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of increase perirenal fat thickness in CKD patients with fatty liver disease. Perirenal fat thickness measured by magnetic resonance imaging (MRI) and pelvic abdominal ultrasound (PAUS). | Baseline
  Correlation between perirenal fat thickness measured by MRI and PAUS and the main markers of kidney function, such as estimated glomerular filtration rate (eGFR), albuminuria and serum urate in CKD patient with FLD.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kamal Abdul_Hamid, prof, Study Director — professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Targher G, Byrne CD. Non-alcoholic fatty liver disease: an emerging driving force in chronic kidney disease. Nat Rev Nephrol. 2017 May;13(5):297-310. doi: 10.1038/nrneph.2017.16. Epub 2017 Feb 20. PMID 28218263
- [Background] Zhang QH, Xie LH, Zhang HN, Liu JH, Zhao Y, Chen LH, Ju Y, Chen AL, Wang N, Song QW, Xie LZ, Liu AL. Magnetic Resonance Imaging Assessment of Abdominal Ectopic Fat Deposition in Correlation With Cardiometabolic Risk Factors. Front Endocrinol (Lausanne). 2022 Mar 30;13:820023. doi: 10.3389/fendo.2022.820023. eCollection 2022. PMID 35432188
- [Background] Wahba IM, Mak RH. Obesity and obesity-initiated metabolic syndrome: mechanistic links to chronic kidney disease. Clin J Am Soc Nephrol. 2007 May;2(3):550-62. doi: 10.2215/CJN.04071206. Epub 2007 Mar 14. PMID 17699463
- [Background] Stenvinkel P, Zoccali C, Ikizler TA. Obesity in CKD--what should nephrologists know? J Am Soc Nephrol. 2013 Nov;24(11):1727-36. doi: 10.1681/ASN.2013040330. Epub 2013 Oct 10. PMID 24115475
- [Background] Chen J, Muntner P, Hamm LL, Jones DW, Batuman V, Fonseca V, Whelton PK, He J. The metabolic syndrome and chronic kidney disease in U.S. adults. Ann Intern Med. 2004 Feb 3;140(3):167-74. doi: 10.7326/0003-4819-140-3-200402030-00007. PMID 14757614
- [Background] Sanches FM, Avesani CM, Kamimura MA, Lemos MM, Axelsson J, Vasselai P, Draibe SA, Cuppari L. Waist circumference and visceral fat in CKD: a cross-sectional study. Am J Kidney Dis. 2008 Jul;52(1):66-73. doi: 10.1053/j.ajkd.2008.02.004. Epub 2008 Apr 28. PMID 18440683
- [Background] Levin A, Stevens PE. Early detection of CKD: the benefits, limitations and effects on prognosis. Nat Rev Nephrol. 2011 Jun 28;7(8):446-57. doi: 10.1038/nrneph.2011.86. PMID 21712852
- [Background] Tonelli M, Dickinson JA. Early Detection of CKD: Implications for Low-Income, Middle-Income, and High-Income Countries. J Am Soc Nephrol. 2020 Sep;31(9):1931-1940. doi: 10.1681/ASN.2020030277. Epub 2020 Aug 24. PMID 32839279
- [Background] Ajmera V, Loomba R. Imaging biomarkers of NAFLD, NASH, and fibrosis. Mol Metab. 2021 Aug;50:101167. doi: 10.1016/j.molmet.2021.101167. Epub 2021 Jan 15. PMID 33460786
- [Background] Byrne CD, Targher G. NAFLD: a multisystem disease. J Hepatol. 2015 Apr;62(1 Suppl):S47-64. doi: 10.1016/j.jhep.2014.12.012. PMID 25920090